CLINICAL TRIAL: NCT07020884
Title: A Randomized, Double-Blind, Placebo-Controlled Phase II Clinical Study to Evaluate the Efficacy, Safety, and Pharmacokinetic Characteristics of ZT002 Injection in Subjects With Overweight or Obesity
Brief Title: A Study of ZT002 Injection With Subjects With Overweight or Obesity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing QL Biopharmaceutical Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BJQL-ZT002-2001
Record Dates: First submitted 2025-06-06; First posted 2025-06-13 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Overweight or Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- ZT002 Injection dose 1 (Experimental): Dose 1 administered subcutaneously (SC), Q2W
  Interventions: Drug: ZT002 Injection
- ZT002 Injection dose 2 (Experimental): Dose 2 administered subcutaneously (SC),Q2W
  Interventions: Drug: ZT002 Injection
- ZT002 Injection dose 3 (Experimental): Dose 3 administered subcutaneously (SC),Q4W
  Interventions: Drug: ZT002 Injection
- ZT002 Injection dose 4 (Experimental): Dose 4 administered subcutaneously (SC), Q4W
  Interventions: Drug: ZT002 Injection
- ZT002 Placebo (Placebo Comparator): administered subcutaneously (SC), Q2W or Q4W
  Interventions: Drug: ZT002 Placebo

INTERVENTIONS:
Drug: ZT002 Injection — Administered SC
  Arms: ZT002 Injection dose 1; ZT002 Injection dose 2; ZT002 Injection dose 3; ZT002 Injection dose 4
Drug: ZT002 Placebo — Administered SC
  Arms: ZT002 Placebo

SUMMARY:
This study will evaluate the percentage change from baseline in weight after 24 weeks of treatment with ZT002 Injection in subjects with overweight/obesity.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and ≤ 75 years.
* BMI ≥28 kg/m², or 24 kg/m2 ≤ BMI < 28 kg/m2 with at least one comorbidity (pre-diabetes, hypertension, hyperlipidemia, fatty liver, obstructive sleep apnoea syndrome due to overweight, weight-bearing joint pain, etc.)
* Weight change is not more than 5% with diet and exercise control alone within 3 months prior to screening.

Exclusion Criteria:

* Previous diagnosis of diabetes; or HbA1c ≥ 6. 5% or fasting blood glucose ≥ 7.0 mmol/L at screening.
* Have used medicines or treatments that affect weight within 3 months prior to screening.
* History of acute or chronic pancreatitis.
* Personal or family (parents, children, and siblings) history of medullary thyroid cancer (MTC) or multiple endocrine neoplasia type II (MEN2).
* History of definite mental disease within 2 years prior to screening or prior suicidal tendency or suicidal behavir; or PHQ-9 scale score is ≥ 15 at screening; or C-SSRS questionnaire is either class 4 or 5 at screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2024-08-14 (Actual); Primary Completion 2025-05-07 (Actual); Study Completion 2025-05-29 (Actual)

PRIMARY OUTCOMES:
The percentage change from baseline in weight after 24 weeks of treatment. | baseline, 24 weeks

SECONDARY OUTCOMES:
The proportion of subjects with weight loss of ≥ 5%, ≥ 10%, and ≥ 15% from baseline after 24 weeks of treatment; | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Linong Ji, MD, Principal Investigator — Peking University People's Hospital
Locations (16):
- China (16):
  - Handan First Hospital, Handan, Hebei
  - Hebei Petro China Cental Hospital, Langfang, Hebei
  - First Hospital of Qinhuangdao, Qinhuangdao, Hebei
  - The Fourth Affiliated Hospital Harbin Medical University, Harbin, Heilongjiang
  - The First Affiliated Hospital of Henan University of Science & Technology, Luoyang, Henan
  - Luoyang Third People's Hospital, Luoyang, Henan
  - The First Affiliated of Nanyang Medical College, Nanyang, Henan
  - Nanjing Jiangning Hospital, Nanjing, Jiangsu
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - Tonghua Central Hospital, Tonghua, Jilin
  - Genertec Liaoyou Gem Flower Hospital, Panjin, Liaoning
  - Central Hospital Affiliated to Shandong First Medical University, Jinan, Shandong
  - Zibo Municipal Hospital, Zibo, Shandong
  - Xi'an Daxing Hospital, Xi’an, Shanxi
  - Peking University First Hospital, Beijing
  - Peking University People's Hospital, Beijing